CLINICAL TRIAL: NCT05466513
Title: Effect of Tactile Stimulation of Facial Skin on Hamstring Flexibility in Healthy Young Males
Brief Title: Facial Tactile Stimulation and Hamstring Flexibility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Masood Khan, Principal Investigator, King Saud University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: RRC-2013-013
Record Dates: First submitted 2022-07-17; First posted 2022-07-20 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Hamstring Flexibility
Keywords: Facial skin; hamstring muscle flexibility; tactile Stimulation

STUDY DESIGN:
Intervention Model Description: Two arms parallel (Experimental and control group) design.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Facial tactile stimulation was applied for 2 minutes.
  Interventions: Other: Facial tactile stimulation
- Control Group (No Intervention): No intervention was applied.

INTERVENTIONS:
Other: Facial tactile stimulation — Tactile stimulation was given around the face with soft tissue paper for two minutes.
  Arms: Experimental Group

SUMMARY:
Inhibition of the sub-occipital muscle group is shown to increase the elasticity of Hamstring muscles. Reversely, stretching of the hamstring muscles is shown to change the pressure pain thresholds over the masseter and upper trapezius muscles. There appears to be a functional link between the neuromuscular system of the head and neck and lower extremities. The present study aimed to investigate the effect of tactile stimulation of facial skin on hamstring length in healthy young males. A total of sixty-six participants participated in the study. Hamstring length was measured by the 'Sit and reach' test in long sitting and 'Toe touch' test in standing position before and after two minutes of facial tactile stimulation in the experimental group and rest in the control group.

DETAILED DESCRIPTION:
Sixty-six young healthy males in the age range 20-30 years participated in the study. They were free of any musculoskeletal conditions that would affect their performance during the test procedures. Subjects were randomly divided into two groups, the experimental group (EG) and control CG) groups. After each subject was briefed about the objectives and procedure of the experiment, written informed consent was obtained. The study fully complied with the ethical standards for human research of our university review board.

The 'Sit and Reach' (SR) test in long sitting and the 'Toe touch' (TT) test in standing were performed according to previously described protocols. Before the start of each testing session of flexibility tests (SR and TT), subjects were asked to perform about 3-5 minutes of warm-up and standardized static stretching exercises focused on the lower back and hamstring muscles.

For the SR test, a strong cubic wooden box of 35 cm was placed against the wall and each subject sat on the floor mat in a long sitting position. The knees were in full extension and the soles of the shoeless feet in neutral ankle position were placed against the box. Subjects were asked to slowly reach forward towards the toes as far as possible while keeping elbows and fingers fully extended, with palms facing down. The subjects had to maintain this position for about five seconds. The distance (in centimeters) between the tips of the middle finger and a reference point on the wooden box was noted.

For the TT test, subjects had to stand upright on the wooden box with feet at hip-width apart and were instructed to bend slowly to reach towards the toes as far as possible while keeping the knees, elbows, and fingers fully extended, with palms facing backward. The subjects had to maintain this position for about five seconds. Again, the distance (in centimeters) between the tips of the middle finger and a reference point on the floor was noted.

For both the SR and the TT tests, the calculated mean recorded distance between the tips of the middle fingers and the reference point during three trials with two-minute rest intervals in-between was used as a reference value for each subject for subsequent analyzes. These mean values were termed Pretest-SR and Pretest TT, respectively. Following the baseline assessment value of the SR and TT tests, each subject of CG or EG underwent three additional trials for each test, with a two-minute interval in between the trials. SR and TT tests were performed randomly without any specific order for both groups of subjects at the same time of day and room temperature. During the two-minute interval, the CG subjects spent their time resting in the supine position with closed eyes, while the EG subjects received tactile stimulation on the facial skin in the supine position with closed eyes. The tactile stimulation to the facial skin of the EG subjects was given by one of the authors and consisted of random strokes similar to a paintbrush around the face with soft tissue paper for two minutes.

For each subject of the CG and EG, the mean distance values between the tips of the middle fingers and the reference point during three trials during the SR and TT tests were calculated, respectively. These mean values were termed Post-test-SR and Post-test-TT, respectively. For all subjects of both the CG and EG, the difference between the Post-test-SR and Pre-test-SR; and Pre-test-TT and Pre-test-TT mean values were calculated. A greater difference between the Post-test-SR and Pre-test-SR; and the Post-test-TT and Pre-test-TT mean values were considered as increased flexibility of the hamstring muscles.

ELIGIBILITY:
Inclusion Criteria:

* young healthy adults

Exclusion Criteria:

* Musculoskeletal disease that can affect the testing.

Ages: 20 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2013-10-10 (Actual); Primary Completion 2014-01-21 (Actual); Study Completion 2014-03-13 (Actual)

PRIMARY OUTCOMES:
Hamstring flexibility | 2 minutes.
  Hamstring muscle length was measured by Sit and reach test and Toe-touch test.

CONTACTS AND LOCATIONS:
Overall Officials: Masood Khan, M.P.Th, Principal Investigator — King Saud University

IPD SHARING:
Plan to Share IPD: No